CLINICAL TRIAL: NCT05761119
Title: Feasibility of an Early Initiated Physiotherapy Intervention Among Patients With Deep Vein Thrombosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, Professor, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-22017283 / 2.1
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Initiated Physiotherapy Intervention (Experimental): All participants will recieve the intervention (see Intervention for description) to investigate the feasibility.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — The focus of the intervention is on exercises that can improve venous return, and consists of progressive walking training at moderate and high intensity as well as guidance on physical activity. The training program is inspired by the WHO's recommendations for physical activity. The training program consists of a 14-day introductory period based on an initial interview with a physiotherapist, where the aim is to hit 30 min. times/day at moderate intensity. After 14 days, the patient receives physiotherapeutic guidance in physical activity and is introduced to the next period of 14 days, where the activity level is maintained, and the goal is to further achieve 2 x 20 min./week of high-intensity physical activity. After one month of training, the patient will be guided on maintaining and possibly progressing physical activity.

SUMMARY:
The project will investigate the feasibility of a physiotherapy intervention for patients diagnosed with deep vein thrombosis for whom a physiotherapy intervention is not currently part of clinical practice in Denmark. Specifically, the project will investigate if an early-initiated physiotherapy intervention for patients who are admitted acutely with first-time deep vein thrombosis (DVT), can be carried out and is experienced as valuable for the patients.

DETAILED DESCRIPTION:
This study aims to investigate whether it is possible for patients diagnosed with DVT to complete early mobilization combined with progressive walking during their hospitalization and the first month after discharge.

This study is twofold. Part one is a clinical cohort study and will investigate the feasibility using quantitative outcomes. Part two is a qualitative study using interviews to investigate the patients' experiences with and attititudes towards a physiotherapy guided intervention of early mobilization combined with progressive walking during their hospitalization and one month after discharge to their own home.

If the physiotherapy intervention is deemed feasible and acceptable, a future randomized controlled trial will investigate the effect of the intervention on quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or above
2. First time lower extremity DVT
3. Hospitalized at the Emergency Department

Exclusion Criteria:

1. Patients without a Danish social security number
2. Terminal patients
3. Patients who do not understand or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Participation | Baseline to one month
  That 50% of all eligible patients wish to participate
Dropout | Baseline to one month
  That less than 20% of the included patients wish to stop the intervention within the first month
Respond rate regarding questionnaire on quality of life | Baseline to one month
  That 80% respond to the questionnaire on quality of life upon admission
Adverse events | Baseline to one month
  That no adverse events, which can be related to the intervention, are recorded during the training period

CONTACTS AND LOCATIONS:
Overall Officials: Helle Juul-Larsen, Ph.D, Principal Investigator — Hvidovre University Hospital; Mette Merete Pedersen, Ph.D, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre, Capital Region
  - Department of Physiotherapy, Næstved-Slagelse-Ringsted Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No